CLINICAL TRIAL: NCT00461331
Title: A Comparison of the Efficacy Beyond 48 Hours of Insulin Aspart (Novolog) and Lispro (Humalog) in Insulin Pumps
Brief Title: Comparison of Insulins Aspart and Lispro in Insulin Pumps
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University Health Sciences Center (Other)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F-0215
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; Glycemic control; Continuous subcutaneous insulin infusion; Continuous glucose monitoring system
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin 1 (Active Comparator): Either insulin Aspart or insulin Lispro were randomized to be insulin 1.
  Interventions: Drug: Insulin Aspart
- Insulin 2 (Active Comparator): Between insulin Aspart and insulin Lispro, the one that was not used as insulin 1 was then used as the second insulin for the second arm of the study.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Aspart — Either one of these insulins were given to the patient as the second insulin (depending on which was given as the first one, the other insulin was insulin 2). Patients used this insulin in the same dose as they did prior to entering the study.
  Other Names: Insulin lispro - insulin Humalog; Insulin aspart - insulin Novolog
  Arms: Insulin 1
Drug: Insulin Lispro — Patients were given either insulin Aspart or Lispro in test period 1. Then they were switched to the other insulin in test period 2.
  Other Names: Insulin Aspart
  Arms: Insulin 2

SUMMARY:
The purpose of the study is to compare the glycemic control between insulins aspart and lispro 48 to 100 hours after pump infusion line change in subjects with type 1 using diabetes using an insulin pump.

DETAILED DESCRIPTION:
Continuous subcutaneous insulin infusion (Insulin pump therapy) is a well established tool for the management of type 1 diabetes. In clinical trials, insulin pump therapy has been shown to have increased efficacy over multiple daily injections. However, the overall glycemic control in patients using insulin pumps has been disappointing. The recommended duration of "needle use" in insulin pump treatment is 48 hours, based on anecdotal observations.

One of the reasons for the suboptimal control may be that patients do not adhere to the advice of changing their pump infusion line every 48 hours. However, it is possible that the loss of glycemic control may be related to instability of insulin in the pump/line. In addition to premeal loss of control after 48 hours of line change, very little is known about post-prandial hyperglycemia leading to loss of efficacy of the insulin via an insulin pump bolus. The development of continuous glucose monitoring system (CGMS) and new tests for short term fluctuations in glucose control such as 1,5-anhydroglucitol make it easier to evaluate the impact of short term loss of control in patients using the insulin pump who delay changing their lines.

The different variables will be compared between the two insulins using a paired t test.

1. Glycemic control will be will be compared 24 to 100 hours after pump infusion line change using CGMS and daily serum 1,5-anhydroglucitol.
2. Post prandial glycemic excursions in plasma glucose following a standardized breakfast 48, 72, and 96 hours after a pump infusion line change will be compared.
3. The used pump infusion line will be collected from the patient and analyzed for insulin binding to the plastic, as well as other possible effects that may determine its role in loss of glycemic control.
4. Comparison of some of the markers of coagulation, inflammation, protein glycation and oxidative stress 48, 72, and 96 hours after a pump infusion line change.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes treated with a pump for at least 3 months

Exclusion Criteria:

* Pregnancy
* Plasma Creatinine > 1.2 mg/dl
* Inability to give informed consent
* HbA1c > 8%
* Known or suspected hypersensitivity to trial drugs or any of their components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-10; Primary Completion 2007-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian A Fonseca, MD, FRCP, Principal Investigator — Tulane Universtiy Health Sciences Center
Locations (1):
- Clinical Translational Unit - Tulane School of Medicine, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Type I diabetes mellitus using an insulin pump were recruited from the outpatient clinics.
Pre-assignment Details: There was no run -in or transition before starting the test period. However, there was a wash out period of up to 2 weeks between the 2 test periods.
Groups:
- Aspart First, Washout, Then Lispro: Patients used Aspart Insulin for up to 100 hours, then entered a two week wash out period, then used Lispro insulin for up to 100 hours. Patients used the insulin at the same dose that they were using prior to entering the study.
- Lispro First, Washout, Then Aspart: Patients used Lispro Insulin for up to 100 hours, then entered a two week wash out period, then used Aspart insulin for up to 100 hours. Patients used the insulin at the same dose that they were using prior to entering the study.
Period: Intervention 1
Arm/Group | Aspart First, Washout, Then Lispro | Lispro First, Washout, Then Aspart
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout
Arm/Group | Aspart First, Washout, Then Lispro | Lispro First, Washout, Then Aspart
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Intervention 2
Arm/Group | Aspart First, Washout, Then Lispro | Lispro First, Washout, Then Aspart
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: These are the characteristics of the entire study population.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Glycemic Control (Glucose Levels Between 180-300 mg/dL) 24 to 100 Hours After Line Change
Description: For each test period, we measured the duration of time that the same pump infusion line could be kept in place without losing glycemic control. Loss of glycemic control was defined as capillary blood glucose level >300 mg/dL.
Time Frame: 24 to 100 hours after last pump infusion line change
Population: The analysis was per protocol, intention to treat. Post-study, glucose readings were grouped according to insulin type and patients ability to maintain Glycemic control(maintaing a glucose level between 180 to 300 mg/dL 24 to 100 hrs after last pump infusion line change)was analyzed for that particular insulin.
Measure: Number; unit: Participants
Groups:
- Insulin Aspart: Patients were randomized to either insulin aspart or lispro in test period 1. They used that insulin for upto 100 hours and then switched to the other insulin after a wash out period of up to 2 weeks. Patients used the insulin at the same dose that they were using prior to entering the study. Post-study, glucose readings were grouped according to insulin type and patients ability to maintain Glycemic control(maintaing a glucose level between 180 to 300 mg/dL 24 to 100 hrs after last pump infusion line change)was analyzed for that particular insulin, in this arm- Aspart.
- Insulin Lispro: Patients were randomized to either insulin aspart or lispro first in test period 1. They used that insulin for upto 100 hours and then switched to the other insulin after a wash out period of up to 2 weeks. Patients used the insulin at the same dose that they were using prior to entering the study. Post-study, glucose readings were grouped according to insulin type and patients ability to maintain Glycemic control(maintaing a glucose level between 180 to 300 mg/dL 24 to 100 hrs after last pump infusion line change)was analyzed for that particular insulin, in this arm- Lispro.
Arm/Group | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 20 | 20
Participants | 17 | 16
Statistical Analysis 1: Comparison: Insulin Aspart vs Insulin Lispro; Glucose levels for patients when they were on each insulin were analyzed. All data was analyzed on an intention to treat basis. Repeated measures, paired t-test and Pearson's correlation on SPSS 14.0 for windows and statistical R-package were used to compare the various variables. This was a pilot study; Test type: Superiority or Other; p = 0.52, Regression, Linear; 7 patients underwent early termination of either one or both of their test period due to loss of glycemic control; Mean Difference (Final Values) = 96.4, 95% CI [87.9 to 100.0], Standard Deviation 8.5

2. Secondary Outcome: Daily Serum Glycomark Levels 48 to 100 Hours After Keeping the Same Pump Infusion Line in Place
Description: Daily serum glycomark levels between day 3 and day 5 after the pump infusion line change. These levels were measured for both the test periods.
Time Frame: 48 to 100 hours after keeping the same pump infusion line in place
Measure: Mean (Standard Deviation); unit: µg/ml
Groups:
- Insulin Lispro: Patients were randomized to either insulin aspart or lispro in test period 1. They used that insulin for upto 100 hours and then switched to the other insulin after a wash out period of up to 2 weeks. Patients used the insulin at the same dose that they were using prior to entering the study. Post-study, glucose readings were grouped according to insulin type and patients ability to maintain Glycemic control(maintaing a glucose level between 180 to 300 mg/dL 24 to 100 hrs after last pump infusion line change)was analyzed for that particular insulin, in this arm- Lispro.
Arm/Group | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 20 | 20
µg/ml | 5.1 (4.13) | 5.6 (4.2)
Statistical Analysis 1: Comparison: Insulin Aspart vs Insulin Lispro; All data was analyzed on an intention to treat basis. Repeated measures, paired t-test and Pearson's correlation on SPSS 14.0 for windows and statistical R-package were used to compare the various variables; Test type: Superiority or Other; p = 0.15, Regression, Linear; Mean Difference (Net) = 5.35, 95% CI [0.97 to 9.23], Standard Deviation 4.165 — This was between days 3 and 5 after the last pump infusion line change using Insulin Aspart and Insulin Lispro. Adequate samples were not available to do the analysis for day 2

3. Secondary Outcome: Oxidative Stress Marker 48, 72 and 96 Hours After Keeping the Same Pump Infusion Line in Place
Description: Free 15-F2t isoprostane was measured between days 3 and 5 after the keeping the same pump infusion line in place. It is a marker of oxidative stress due to hyperglycemia that was being compared between the two test periods.
Time Frame: Between 48, 72 and 96 hours after the last pump infusion line change
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Insulin Aspart | Insulin Lispro
Number analyzed (Participants) | 20 | 20
pg/ml | 6.9 (2.5) | 6.5 (2.2)
Statistical Analysis 1: Comparison: Insulin Aspart vs Insulin Lispro; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.55, Regression, Linear; Mean Difference (Net) = 6.7, 95% CI [4.4 to 9.4], Standard Deviation 2.35 — This was for test period 1 between days 3 and 5 after the last pump infusion line change

ADVERSE EVENTS:
Arm/Group | Insulin Aspart | Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No